CLINICAL TRIAL: NCT03101137
Title: Effects Of Adjuvants (Dexamethasone and Dexmedetomidine) to Caudal Anesthesia on Cardiac Output and Hemodynamics Measured By Electrical Cardiometry In Children: A Randomized Double Blind Study
Brief Title: Effects Of Adjuvants to Caudal Anesthesia on Hemodynamics Measured By Electrical Cardiometry In Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Doaa Fawzy Abd El Fattah Hassan, Assistant lecturer of anesthesia, surgical ICU and pain management - Cairo University, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N6-2016/MD
Record Dates: First submitted 2016-11-14; First posted 2017-04-04 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Caudal Block
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Caudal block with dexmedetomedine (Active Comparator): Caudal Dexmedetomidine block group (DEXM) (n= 16) will receive caudal block using the bupivacaine 0.25% and Dexmedetomidine 1 μg/kg with the conventional general anesthesia,
  Interventions: Drug: Caudal block with dexmedetomedine
- Caudal block with dexamethasone (Active Comparator): caudal Dexamethasone Block group (DEXA) (n =16) will receive caudal block using the bupivacaine 0.25% and Dexamethasone 0.1 mg/kg with the conventional general anesthesia,
  Interventions: Drug: Caudal dexamethasone
- Control (caudal block with bupivacaine) (Placebo Comparator): caudal with bubivacaine (CONTROL) group (n = 16) will receive caudal block using the bupivacaine 0.25% and general anesthesia.
  Interventions: Drug: Control (bupivacaine)

INTERVENTIONS:
Drug: Caudal block with dexmedetomedine — After induction, the electrical cardiometry is applied in supine position and a measurement for the baseline cardiac output, systemic vascular resistance and stroke volume is taken. In left lateral position, the back is sterilized. The block is done by introducing a 23-gauge needle perpendicular to the sacrococcygeal membrane. The needle is inserted until there is release of resistance as it pierces the sacro-coccygeal membrane. Then, it is directed upwards to make an angle of 20-30° with the skin about 2 mm. 1 ml/kg bupivacaine 0.25% along with dexmedetomidine 1 μg/kg (diluted with normal saline to 1ml) is injected over about 60s. Then, another measurement for the hemodynamics is taken at 5, 10, 20 and 30 minutes after caudal block.
  Other Names: Precedex
  Arms: Caudal block with dexmedetomedine
Drug: Caudal dexamethasone — After induction, the electrical cardiometry is applied in supine position and a measurement for the baseline cardiac output, systemic vascular resistance and stroke volume is taken. In left lateral position, the back is sterilized. The block is done by introducing a 23-gauge needle perpendicular to the sacrococcygeal membrane. The needle is inserted until there is release of resistance as it pierces the sacro-coccygeal membrane. Then, it is directed upwards to make an angle of 20-30° with the skin about 2 mm. 1 ml/kg bupivacaine 0.25% along with dexamethasone 0.1mg/kg (diluted with normal saline to 1ml) is injected over about 60s. Then, another measurement for the hemodynamics is taken at 5, 10, 20 and 30 minutes after caudal block.
  Other Names: Decadrone
  Arms: Caudal block with dexamethasone
Drug: Control (bupivacaine) — After induction, the electrical cardiometry is applied in supine position and a measurement for the baseline cardiac output, systemic vascular resistance and stroke volume is taken. In left lateral position, the back is sterilized. The block is done by introducing a 23-gauge hypodermic needle perpendicular to the sacrococcygeal membrane. The needle is inserted until there is release of resistance as it pierces the sacro-coccygeal membrane. Then, it is directed upwards to make an angle of 20-30° with the skin about 2 mm. 1 ml/kg the control (bupivacaine) 0.25% is injected over about 60s. Then, another measurement for the hemodynamics is taken at 5, 10, 20 and 30 minutes after caudal block.
  Other Names: Marcaine
  Arms: Control (caudal block with bupivacaine)

SUMMARY:
Caudal epidural anesthesia is one of the most common regional techniques used for post-operative pain management in pediatric patients. In this study we are going to compare the effects of caudal bupivacaine , caudal Dexamethasone with bubivacaine and Dexmedetomidine with bupivacaine on the systemic vascular resistance and the cardiac output, in pediatric patients undergoing lower abdominal surgeries, by using the electrical cardiometry (EC).

DETAILED DESCRIPTION:
Participants will be randomly allocated by a computer-generated table into one of the 3 study groups; the randomization sequence was concealed in sealed envelopes. The three study groups were as follows:

Group A: Caudal Dexmedetomidine block group (DEXM) (n= 16) will receive caudal block using the bupivacaine 0.25% and Dexmedetomidine 1 μg/kg with the conventional general anesthesia,

Group B: caudal Dexamethasone Block group (DEXA) (n =16) will receive caudal block using the bupivacaine 0.25% and Dexamethasone 0.1 mg/kg with the conventional general anesthesia,

Group C: caudal with bubivacaine (CONTROL) group (n = 16) will receive caudal block using the bupivacaine 0.25% and general anesthesia.

After induction of general anesthesia, the electrodes of the electrical cardiometry will be applied on the child neck and chest in the supine position and a measurement for the baseline cardiac output, systemic vascular resistance and stroke volume will be taken using the electrical cardiometry. Baseline blood pressure and heart rate will be also recorded.Then, another measurement for the systemic cardiac output, vascular resistance, stroke volume heart rate and blood pressure will be taken at 5minutes, 10 minutes, 20 minutes and 30 minutes after caudal block. The measurements will be stored and analyzed off-line.

The Electrical Cardiometry device that will be used is the ICON™ monitor; (the Portable Noninvasive Hemodynamic Monitor manufactured by Osypka Medical Company). The measurements will be stored and analyzed off-line. The average values during three consecutive measures will be considered for the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients 1 - 7 years.
2. Both genders (male & female).
3. ASA I & ASA II patients.
4. Children scheduled for lower abdominal elective surgeries including genitourinary and perineal regions surgeries.

Exclusion Criteria:

1. Parents' refusal of regional block.
2. Patients requiring emergency procedures.
3. Bleeding disorders.
4. Skin lesions or wounds at site of proposed needle insertion.
5. Cutaneous anomalies (angioma, hair tuft, nevus or a dimple) near the puncture point requiring radiological examination (ultrasound, CT or MRI).
6. Progressive neurological disorders.
7. Patients with congenital heart disease.
8. Patients with Allergies to used drugs
9. Surgeries with large fluid shift or massive blood loss.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac output | up to 30 minutes
  Cardiac output at 5 minutes, 10 minutes, 20 minutes and 30 minutes after caudal block,the cardiac output is measured with L/minute

CONTACTS AND LOCATIONS:
Overall Officials: Nevine M Gouda, professor, Study Chair — Kasr El Aini Hospitals-Cairo university-Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1) Shah N., Patel J., Chhaya A. and Upadhyaya R. Comparison of general anesthesia v/s caudal epidural in pediatric infra umbilical surgeries. International J of Biomed Res. 2015; 6(01): 35- 9.
- [Background] 2) Almajali Z., Batarseh E., Daameh S., Qabha A. and Haddadin M. Comparison of Postoperative Pain Relief Impact between Caudal Bupivacaine Alone and Caudal Bupivacaine-Dexamethasone Mixture Administration for Pediatric Local Tube Urethroplasty. J of The R Med Serv. 2014; 21(4): 19-24.
- [Background] 3) Butterworth J., Mackey,D. & Wasnick,J. Morgan & Mikhail's Clinical Anesthesiology. 5th ed. the United States: McGraw-Hill Education, LLC. 2013; 877-905.
- [Background] Farrag WS, Ibrahim AS, Mostafa MG, Kurkar A, Elderwy AA. Ketamine versus magnesium sulfate with caudal bupivacaine block in pediatric inguinoscrotal surgery: A prospective randomized observer-blinded study. Urol Ann. 2015 Jul-Sep;7(3):325-9. doi: 10.4103/0974-7796.152039. PMID 26229319
- [Background] 5) Bhaskar D. , Kumar P. , Mridul S. , Vipin D. , Vivek T. and Mohamed A. Comparison Of Caudal Dexmedetomidine And Fentanyl For Postoperative Analgesia. J of Adv Res in Bio Scien. 2014; 6 (1) 51-7.
- [Background] 6) El Gendy H.A. & Elsharnouby N.M. Ultrasound Guided Single Injection Caudal Epidural Anesthesia Of Isobaric Bupivacaine With/Without Dexamethasone For Geriatric Patients Undergoing Total Hip Replacement Surgery. Egyptian Journal of Anesthesia. 2014; 30: 293- 8.
- [Background] Deng M, Wang X, Wang L, Zheng S. The hemodynamic effects of newborn caudal anesthesia assessed by transthoracic echocardiography: a randomized, double-blind, controlled study. Paediatr Anaesth. 2008 Nov;18(11):1075-81. doi: 10.1111/j.1460-9592.2008.02786.x. PMID 18950332
- [Background] Galante D, Pellico G, Meola S, Caso A, De Capraris A, Milillo R, Mirabile C, Olivieri M, Cinnella G, Dambrosio M. Hemodynamic effects of levobupivacaine after pediatric caudal anesthesia evaluated by transesophageal doppler. Paediatr Anaesth. 2008 Nov;18(11):1066-74. doi: 10.1111/j.1460-9592.2008.02774.x. PMID 18950331
- [Background] Larousse E, Asehnoune K, Dartayet B, Albaladejo P, Dubousset AM, Gauthier F, Benhamou D. The hemodynamic effects of pediatric caudal anesthesia assessed by esophageal Doppler. Anesth Analg. 2002 May;94(5):1165-8, table of contents. doi: 10.1097/00000539-200205000-00020. PMID 11973181
- [Background] 10) Rajput RS, Das S., Chauhan S., Bisoi AK. & Vasdev S. Comparison of Cardiac Output Measurement by Noninvasive Method with Electrical Cardiometry and Invasive Method with Thermodilution Technique in Patients Undergoing Coronary Artery Bypass Grafting. Wor J Cardiovas S. 2014 ;(4): 123-130.
- [Background] Xiang Q, Huang DY, Zhao YL, Wang GH, Liu YX, Zhong L, Luo T. Caudal dexmedetomidine combined with bupivacaine inhibit the response to hernial sac traction in children undergoing inguinal hernia repair. Br J Anaesth. 2013 Mar;110(3):420-4. doi: 10.1093/bja/aes385. Epub 2012 Nov 15. PMID 23161357
- [Background] Mason KP, Lerman J. Review article: Dexmedetomidine in children: current knowledge and future applications. Anesth Analg. 2011 Nov;113(5):1129-42. doi: 10.1213/ANE.0b013e31822b8629. Epub 2011 Aug 4. PMID 21821507
- [Background] 13) Almajali Z., Batarseh E., Daameh S., Qabha A., Haddadin M. Comparison Of Postoperative Pain Relief Impact Between Caudal Bupivacaine Alone And Caudal Bupivacaine-Dexamethasone Mixture Administration For Pediatric Local Tube Urethroplasty. J Roy Med Serv. 2014; 21(4): 19-24.
- [Background] 14) Dalal S., Paul A. and Tirpude NG. Clinical Evaluation of Caudal Clonidine as an Adjuvant to Bupivacaine in Pediatric Patients Undergoing Sub Umbilical Surgeries. Research Chronicle in health sciences. 2015; 1(2): 110-121.
- [Background] 15) Alsadek W., Al-Gohari M., Elsonbaty M., Nassar N.& Alkonaiesy R. Ultrasound Guided TAP Block Versus Ultrasound Guided Caudal Block For Pain Relief In Children Undergoing Lower Abdominal Surgeries. Egyp J of Anaesth. 2015; (31): 155-160.